CLINICAL TRIAL: NCT00626990
Title: Phase III Trial on Concurrent and Adjuvant Temozolomide Chemotherapy in Non-1p/19q Deleted Anaplastic Glioma. The CATNON Intergroup Trial.
Brief Title: Phase III Trial of Anaplastic Glioma Without 1p/19q Loss of Heterozygosity (LOH)
Acronym: CATNON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: NCIC Clinical Trials Group (Network); Radiation Therapy Oncology Group (Network); Medical Research Council (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-26053-22054; NCIC CTG CEC.1 (Other: NCI-C); RTOG-0834 (Other: RTOG); 2006-001533-17 (EudraCT Number); P04839 (Other Grant/Funding Number: Merck); MRC BR14 (Other: MRC CTU)
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Results first posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; adult anaplastic astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Astrocytoma | interventions — Temozolomide; DNA Methylation; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Radiotherapy (RT) alone (Active Comparator): radiation therapy alone
  Interventions: Genetic: DNA methylation analysis; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment; Radiation: radiation therapy
- RT & Concurrent CT (Active Comparator): Radiotherapy and concurrent temozolomide chemotherapy
  Interventions: Drug: temozolomide; Genetic: DNA methylation analysis; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment; Radiation: radiation therapy
- RT + Adjuvant CT (Active Comparator): Radiotherapy plus adjuvant temozolomide chemotherapy
  Interventions: Drug: temozolomide; Genetic: DNA methylation analysis; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: quality-of-life assessment; Radiation: radiation therapy
- RT & Concurrent CT + adjuvant CT (Active Comparator): Radiotherapy and concurrent chemotherapy plus adjuvant temozolomide chemotherapy
  Interventions: Drug: temozolomide; Genetic: DNA methylation analysis; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: quality-of-life assessment; Radiation: radiation therapy

INTERVENTIONS:
Drug: temozolomide — Patients randomized to concomitant temozolomide will receive temozolomide continuously at a daily dose of 75 mg/m² during radiotherapy.
  Other Names: Temodar; Temodal
  Arms: RT & Concurrent CT; RT & Concurrent CT + adjuvant CT; RT + Adjuvant CT
Genetic: DNA methylation analysis — O6-Methylguanine-DNA Methyltransferase (MGMT) methylation status is used for stratification at randomization.
Other: laboratory biomarker analysis — Prognostic factor analyses
Procedure: adjuvant therapy — Patients randomized to adjuvant temozolomide will start adjuvant temozolomide after a 4 week resting period after the end of radiotherapy.
  Arms: RT & Concurrent CT + adjuvant CT; RT + Adjuvant CT
Procedure: quality-of-life assessment — Quality of Life analysis will also be used to assess neurological deterioration free progression
Radiation: radiation therapy — Radiotherapy will consist of a conventionally fractionated regimen for 6.5 weeks in a once daily schedule

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with temozolomide may kill more tumor cells. It is not yet known whether giving temozolomide during and/or after radiation therapy is more effective than radiation therapy alone in treating anaplastic glioma.

PURPOSE: This randomized phase III trial is studying giving temozolomide during and/or after radiation therapy to see how well it works compared to radiation therapy alone in treating patients with anaplastic glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether concurrent radiotherapy with daily temozolomide improves overall survival as compared to no daily temozolomide in patients with non-1p/19q deleted anaplastic glioma.
* To assess whether adjuvant temozolomide improves survival as compared to no adjuvant temozolomide in patients with non-1p/19q deleted anaplastic glioma.

Secondary

* To assess whether concurrent and adjuvant temozolomide prolongs progression-free survival and neurological deterioration-free survival in patients with non-1p/19q deleted anaplastic glioma.
* To assess the safety of concurrent and adjuvant temozolomide in patients with non-1p/19q deleted anaplastic glioma, including late effects on cognition.
* To assess the impact of concurrent and adjuvant temozolomide on the quality of life of patients with non-1p/19q deleted anaplastic glioma.

OUTLINE: This is a multicenter study. Patients are stratified according to institution, World Health Organization (WHO) performance status (0 vs > 0), age (≤ 50 vs > 50), presence of 1p LOH only (yes vs no), presence of oligodendroglial elements (yes vs no), and O6-methylguanine-DNA methyltransferase promoter methylation status (methylated vs unmethylated vs indeterminate). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients undergo radiotherapy* once daily, 5 days a week, for 6.5 weeks (total of 33 fractions).
* Arm II: Patients undergo radiotherapy* once daily, 5 days a week and receive oral temozolomide once daily for 6.5 weeks (total of 33 fractions of radiotherapy).
* Arm III: Patients undergo radiotherapy* once daily, 5 days a week for 6.5 weeks (total of 33 fractions). Beginning 4 weeks after completion of radiotherapy, patients receive adjuvant oral temozolomide once daily on days 1-5. Treatment with adjuvant temozolomide repeats every 28 days for up to 12 courses.
* Arm IV: Patients undergo radiotherapy* once daily, 5 days a week and receive oral temozolomide once daily for 6.5 weeks (total of 33 fractions of radiotherapy). Beginning 4 weeks after completion of radiotherapy, patients receive adjuvant oral temozolomide once daily on days 1-5. Treatment with adjuvant temozolomide repeats every 28 days for up to 12 courses.
* Patients must begin radiotherapy within 8 days after randomization and within 7 weeks after surgery.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of-life questionnaires, including EORTC core quality of life questionnaire (QLQ-C30) version 3, EORTC brain cancer module (BCM20), and the Mini Mental Status Exam at baseline, 4 weeks after the completion of radiotherapy, and then every 3 months for 5 years.

Tissue samples are collected at baseline for histology review, 1p/19q analysis, methylation status of the O6-methylguanine-DNA methyltransferase promoter, and isocitrate dehydrogenase mutation analysis.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Anaplastic oligodendroglioma
  * Anaplastic oligoastrocytoma
  * Anaplastic astrocytoma
* Newly diagnosed disease
* Prior surgery for a low grade tumor is allowed, provided histological confirmation of an anaplastic tumor is present at the time of progression
* Absence of combined 1p/19q loss
* Tumor material available for central 1p/19q assessment, central O6-methylguanine-DNA methyltransferase promoter methylation status assessment, isocitrate dehydrogenase mutation analysis, and central pathology review
* Patients must be on a stable or decreasing dose of steroids for at least two weeks prior to randomization

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9 cells/L
* Platelet count ≥ 100 x 10^9 cells/L
* Bilirubin < 1.5 x upper limit of normal (ULN)
* Alkaline phosphatase < 2.5 x ULN
* Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) < 2.5 x ULN
* Serum creatinine < 1.5 x ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known HIV infection or chronic hepatitis B or hepatitis C infection
* No other serious medical condition that would interfere with follow-up
* No medical condition that could interfere with oral medication intake (e.g., frequent vomiting or partial bowel obstruction)
* No other prior malignancies except for any malignancy which was treated with curative intent more than 5 years prior to registration and adequately controlled limited basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix
* No prior or concurrent malignancies at other sites except for surgically cured carcinoma in situ of the cervix or nonmelanoma skin cancer
* No psychological, familial, sociological, or geographical condition that would potentially hamper compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, including carmustine-containing wafers (Gliadel®)
* No prior radiotherapy to the brain
* No concurrent growth factors unless vital for the patient
* No other concurrent investigational treatment
* No other concurrent anticancer agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2029-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, Study Chair — Universitatsklinikum Heidelberg; Warren P. Mason, MD, Study Chair — Princess Margaret Hospital, Canada; Michael A. Vogelbaum, MD, PhD, Study Chair — The Cleveland Clinic; S. Erridge, Study Chair — Medical Research Council; Anna Nowak, MD, Study Chair — Sir Charles Gairdner Hospital - Nedlands
Locations (132):
- United States (72):
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCSF University of California San Francisco Medical Center-Mount Zion, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital, Fort Wayne, Indiana
  - Saint Vincent Oncology Center, Indianapolis, Indiana
  - McFarland Clinic, Ames, Iowa
  - June E. Nylen Cancer Center, Sioux City, Iowa
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Maine Medical Center, Scarborough, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachussets General Hospital Cancer Center, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - St John's Mercy Medical Center, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - State University of New York Upstate Medical University, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester - James P. Wilmot Cancer Center, Rochester, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Akron City Hospital - Summa Health System, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Western Reserve University, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - UHHS - Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - UPMC - Heritage Valley Health System - The Medical Center, Beaver, Pennsylvania
  - Penn State M.S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Radiation Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - University of Texas Medical Branch, Galveston, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - University Of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran, La Crosse, Wisconsin
  - University Of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Australia (10):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Melbourne Hospital, Parkville, Victoria
  - Flinders Medical Centre, Bedford Park
  - Austin-Repatriation Medical Centre, Heidelberg
  - Royal Hobart Hospital, Hobart
  - St Vincent'S Hospital, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
  - Alfred Hospital, Prahran
- Belgium (6):
  - ZNA Middelheim, Antwerp
  - Cliniques Universitaires St. Luc, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Clinique Notre-Dame, Charleroi
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - U.Z. Gasthuisberg, Leuven
- Canada (5):
  - Tom Baker Cancer Centre, Calgary
  - London Regional Cancer Center, London
  - Allan Blair Cancer Centre, Saskatoon
  - University Health Network - Oci / Princess Margaret Hospital, Toronto
  - Cancercare Manitoba, Winnipeg
- France (6):
  - Assistance Publique - Hôpitaux de Marseille - C.H.U. De La Timone, Marseille
  - C.H.U. de Nancy - Hopital St Julien, Nancy
  - Centre Antoine Lacassagne, Nice
  - Chu Pitie-Salpetriere AP-HP, Paris
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Klinikum Bamberg, Bamberg
  - Universitaetsklinikum Bonn, Bonn
  - Medizinische Hochschule Hannover, Hanover
  - UniversitaetsKlinikum Heidelberg, Heidelberg
  - Universitaetskliniken Regensburg, Regensburg
  - Universitaetsklinikum Tuebingen, Tübingen
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (3):
  - Ospedale Bellaria, Bologna
  - Istituto Scientifico H.S. Raffaele, Milan
  - Azienda Ospedaliera San Giovanni Battista Di Torino-Universita Di Torino, Torino
- Netherlands (7):
  - Academisch Medisch Centrum - Universiteit van Amsterdam, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastro Clinic - Maastricht Radiation Oncology, Maastricht
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Erasmus MC - Daniel den Hoed Cancer Center, Rotterdam
  - Medisch Centrum Haaglanden - Westeinde, The Hague
- Spain (2):
  - Hospital Clinic Universitari, Barcelona
  - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Barcelona
- Switzerland (2):
  - Hopital Cantonal Universitaire De Geneve, Geneva
  - Universitaetsspital, Zurich
- United Kingdom (12):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol
  - Addenbrookes Hospital, Cambridge
  - Cheltenham General Hospital, Cheltenham
  - Western General Hospital, Edinburgh
  - Royal Devon And Exeter Hospital, Exeter
  - St. James'S University Hospital, Leeds
  - Christie NHS Foundation Trust, Manchester
  - Clatterbridge Centre for Oncology NHS Trust, Metropolitan Borough of Wirral
  - Nottingham University Hospitals NHS Trust - City Hospital campus, Nottingham
  - Derriford Hospital, Plymouth
  - Weston Park Hospital, Sheffield
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] van den Bent MJ, Ghisai SA, Wick W, Sanson M, Brandes AA, Clement PM, Erridge SC, Vogelbaum MA, Nowak AK, Baurain JF, Mason WP, Wheeler H, Tabouret E, Gill S, Griffin M, Taal W, Ruda R, Weller M, McBain C, Reijneveld JC, Enting RH, Tran S, Lesimple T, Kocher M, Gijtenbeek A, Lim E, Herrlinger U, Hau P, Dhermain F, Aldape K, Jenkins RB, Dubbink HJ, Kros JM, Wesseling P, Hoogstrate Y, Nuyens S, Golfinopoulos V, Tesileanu CMS, Gorlia T, French P, Baumert BG. Concurrent and adjuvant temozolomide for 1p/19q non-co-deleted anaplastic glioma (CATNON; EORTC study 26053-22054): final and exploratory analyses of a randomised, open-label, phase 3 trial. Lancet Oncol. 2026 Jan;27(1):45-56. doi: 10.1016/S1470-2045(25)00614-X. PMID 41449147
- [Derived] Tesileanu CMS, Sanson M, Wick W, Brandes AA, Clement PM, Erridge SC, Vogelbaum MA, Nowak AK, Baurain JF, Mason WP, Wheeler H, Chinot OL, Gill S, Griffin M, Rogers L, Taal W, Ruda R, Weller M, McBain C, van Linde ME, Aldape K, Jenkins RB, Kros JM, Wesseling P, von Deimling A, Hoogstrate Y, de Heer I, Atmodimedjo PN, Dubbink HJ, Brouwer RWW, van IJcken WFJ, Cheung KJ, Golfinopoulos V, Baumert BG, Gorlia T, French PJ, van den Bent MJ. Temozolomide and Radiotherapy versus Radiotherapy Alone in Patients with Glioblastoma, IDH-wildtype: Post Hoc Analysis of the EORTC Randomized Phase III CATNON Trial. Clin Cancer Res. 2022 Jun 13;28(12):2527-2535. doi: 10.1158/1078-0432.CCR-21-4283. PMID 35275197
- [Derived] van den Bent MJ, Tesileanu CMS, Wick W, Sanson M, Brandes AA, Clement PM, Erridge S, Vogelbaum MA, Nowak AK, Baurain JF, Mason WP, Wheeler H, Chinot OL, Gill S, Griffin M, Rogers L, Taal W, Ruda R, Weller M, McBain C, Reijneveld J, Enting RH, Caparrotti F, Lesimple T, Clenton S, Gijtenbeek A, Lim E, Herrlinger U, Hau P, Dhermain F, de Heer I, Aldape K, Jenkins RB, Dubbink HJ, Kros JM, Wesseling P, Nuyens S, Golfinopoulos V, Gorlia T, French P, Baumert BG. Adjuvant and concurrent temozolomide for 1p/19q non-co-deleted anaplastic glioma (CATNON; EORTC study 26053-22054): second interim analysis of a randomised, open-label, phase 3 study. Lancet Oncol. 2021 Jun;22(6):813-823. doi: 10.1016/S1470-2045(21)00090-5. Epub 2021 May 14. PMID 34000245
- [Derived] van den Bent MJ, Baumert B, Erridge SC, Vogelbaum MA, Nowak AK, Sanson M, Brandes AA, Clement PM, Baurain JF, Mason WP, Wheeler H, Chinot OL, Gill S, Griffin M, Brachman DG, Taal W, Ruda R, Weller M, McBain C, Reijneveld J, Enting RH, Weber DC, Lesimple T, Clenton S, Gijtenbeek A, Pascoe S, Herrlinger U, Hau P, Dhermain F, van Heuvel I, Stupp R, Aldape K, Jenkins RB, Dubbink HJ, Dinjens WNM, Wesseling P, Nuyens S, Golfinopoulos V, Gorlia T, Wick W, Kros JM. Interim results from the CATNON trial (EORTC study 26053-22054) of treatment with concurrent and adjuvant temozolomide for 1p/19q non-co-deleted anaplastic glioma: a phase 3, randomised, open-label intergroup study. Lancet. 2017 Oct 7;390(10103):1645-1653. doi: 10.1016/S0140-6736(17)31442-3. Epub 2017 Aug 8. PMID 28801186
- See also: Clinical trial summary from the EORTC database — https://www.eortc.org/research_field/clinical-detail/26053/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After registration step was completed, eligible patients were randomized into the trial within 8 days from the start of radiotherapy; at this time, all baseline requirements for the study had to be fulfilled.
Pre-assignment Details: The patients were first registered to the trial by authorized sites. For all patients, tumor and blood samples had to be sent for histology review, 1p/19q analysis and O6-Methylguanine-DNA Methyltransferase (MGMT) assay. If inclusion was based on central pathology and 1p/19q diagnosis the patient could be randomized into the trial once found eligible at central assessment.
Groups:
- RT Alone: radiation therapy alone
  DNA methylation analysis: MGMT methylation status is used for stratification at randomization.
  laboratory biomarker analysis: Prognostic factor analyses
  quality-of-life assessment: Quality of Life analysis will also be used to assess neurological deterioration free progression
  radiation therapy: Radiotherapy will consist of a conventionally fractionated regimen for 6.5 weeks in a once daily schedule
- RT & Concurrent CT: Radiotherapy and concurrent temozolomide chemotherapy
  temozolomide: Patients randomized to concomitant temozolomide will receive temozolomide continuously at a daily dose of 75 mg/m² during radiotherapy.
  DNA methylation analysis: MGMT methylation status is used for stratification at randomization.
  laboratory biomarker analysis: Prognostic factor analyses
  quality-of-life assessment: Quality of Life analysis will also be used to assess neurological deterioration free progression
  radiation therapy: Radiotherapy will consist of a conventionally fractionated regimen for 6.5 weeks in a once daily schedule
- RT + Adjuvant CT: Radiotherapy plus adjuvant temozolomide chemotherapy
  temozolomide: Patients randomized to concomitant temozolomide will receive temozolomide continuously at a daily dose of 75 mg/m² during radiotherapy.
  DNA methylation analysis: MGMT methylation status is used for stratification at randomization.
  laboratory biomarker analysis: Prognostic factor analyses
  adjuvant therapy: Patients randomized to adjuvant temozolomide will start adjuvant temozolomide after a 4 week resting period after the end of radiotherapy.
  quality-of-life assessment: Quality of Life analysis will also be used to assess neurological deterioration free progression
  radiation therapy: Radiotherapy will consist of a conventionally fractionated regimen for 6.5 weeks in a once daily schedule
- RT & Concurrent CT + Adjuvant CT: Radiotherapy and concurrent chemotherapy plus adjuvant temozolomide chemotherapy
  temozolomide: Patients randomized to concomitant temozolomide will receive temozolomide continuously at a daily dose of 75 mg/m² during radiotherapy.
  DNA methylation analysis: MGMT methylation status is used for stratification at randomization.
  laboratory biomarker analysis: Prognostic factor analyses
  adjuvant therapy: Patients randomized to adjuvant temozolomide will start adjuvant temozolomide after a 4 week resting period after the end of radiotherapy.
  quality-of-life assessment: Quality of Life analysis will also be used to assess neurological deterioration free progression
  radiation therapy: Radiotherapy will consist of a conventionally fractionated regimen for 6.5 weeks in a once daily schedule
Period: Overall Study
Arm/Group | RT Alone | RT & Concurrent CT | RT + Adjuvant CT | RT & Concurrent CT + Adjuvant CT
Started | 189 | 188 | 186 | 188
Completed | 175 | 163 | 109 | 93
Not Completed | 14 | 25 | 77 | 95
Not completed — Lack of Efficacy | 6 | 7 | 49 | 40
Not completed — Adverse Event | 1 | 7 | 14 | 28
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 5 | 11
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Various different reasons/missing | 4 | 8 | 8 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RT Alone | RT & Concurrent CT | RT + Adjuvant CT | RT & Concurrent CT + Adjuvant CT | Total
Number analyzed (Participants) | 189 | 188 | 186 | 188 | 751
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 174 | 168 | 174 | 180 | 696
  >=65 years | 15 | 20 | 12 | 8 | 55
Age, Continuous [Median (Full Range); unit: years] | 42 [19 to 81.2] | 43.1 [20.1 to 77.1] | 40 [20 to 82.3] | 42.8 [18.3 to 80.1] | 42.2 [18.3 to 82.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 68 | 82 | 82 | 307
  Male | 114 | 120 | 104 | 106 | 444
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 5 | 6 | 6 | 23
  Netherlands | 19 | 20 | 19 | 14 | 72
  Belgium | 19 | 20 | 16 | 18 | 73
  United States | 30 | 22 | 21 | 28 | 101
  Italy | 13 | 10 | 16 | 11 | 50
  United Kingdom | 31 | 39 | 39 | 34 | 143
  Australia | 14 | 22 | 21 | 25 | 82
  France | 26 | 23 | 22 | 22 | 93
  Switzerland | 5 | 7 | 7 | 7 | 26
  Germany | 22 | 13 | 17 | 18 | 70
  Spain | 4 | 6 | 1 | 3 | 14
  Turkey | 0 | 1 | 1 | 2 | 4
Presence of oligodendroglial elements [Count of Participants; unit: Participants]
  No | 146 | 144 | 143 | 144 | 577
  Yes | 43 | 44 | 43 | 44 | 174
World Health Organization (WHO) Performance Status [Count of Participants; unit: Participants]
  ECOG performance status 0 (good prognosis) | 111 | 110 | 108 | 112 | 441
  ECOG performance status >0 (poorer prognosis) | 78 | 78 | 78 | 76 | 310
Procedure for pathology and genetic testing [Count of Participants; unit: Participants]
  by local site laboratory assessment | 70 | 70 | 68 | 54 | 262
  by central laboratory assessment | 119 | 118 | 116 | 134 | 487
  Unknown | 0 | 0 | 2 | 0 | 2
Presence of 1p LOH [Count of Participants; unit: Participants]
  No loss | 175 | 176 | 172 | 175 | 698
  Loss | 14 | 12 | 14 | 13 | 53
MGMT Methylation status [Count of Participants; unit: Participants]
  Methylated | 62 | 55 | 66 | 56 | 239
  Unmethylated | 83 | 79 | 78 | 87 | 327
  Undetermined/invalid | 44 | 54 | 42 | 45 | 185

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival as Measured From the Day of Randomization
Description: The duration of survival is the time interval between randomization and the date of death due to any cause. Patients not reported dead or lost to follow up will be censored at the date of the last follow up examination.
Time Frame: from date from enrollment till the date of death (time till death is up to 10.9 years after patient enrollment in the study)
Population: This trial studied 2 questions 1) effect of concomitant Temozolomide (TMZ) 2) effect of adjuvant TMZ. The 4 randomized arms were combined. Absence of concomitant TMZ including Arm Radiotherapy (RT) alone & Arm RT followed by adjuvant TMZ. Presence of concomitant TMZ including Arm TMZ/RT & Arm TMZ/RT followed by adjuvant TMZ. Absence of adjuvant TMZ including Arm RT alone & Arm TMZ/RT. Presence of adjuvant TMZ including Arm RT followed by adjuvant TMZ & Arm TMZ/RT followed by adjuvant TMZ
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Absence of Concomitant Temozolomide (TMZ): Including 2 randomized arms: Arm RT alone and Arm RT followed by adjuvant TMZ
- Presence of Concomitant Temozolomide (TMZ): Including 2 randomized arms: Arm TMZ/RT and Arm TMZ/RT followed by adjuvant TMZ
- Absence of Adjuvant Temozolomide (TMZ): Including two randomized arms: Arm RT alone and Arm TMZ/RT
- Presence of Adjuvant Temozolomide (TMZ): Including to 2 randomized arms: Arm RT followed by adjuvant TMZ and Arm TMZ/RT followed by adjuvant TMZ
Arm/Group | Absence of Concomitant Temozolomide (TMZ) | Presence of Concomitant Temozolomide (TMZ) | Absence of Adjuvant Temozolomide (TMZ) | Presence of Adjuvant Temozolomide (TMZ)
Number analyzed (Participants) | 375 | 376 | 377 | 374
Months | 60.42 [45.7 to 71.49] | 66.92 [48.53 to 82.33] | 46.92 [37.88 to 56.94] | 82.33 [67.19 to 116.63]
Statistical Analysis 1: Comparison: Absence of Concomitant Temozolomide (TMZ) vs Presence of Concomitant Temozolomide (TMZ); Test type: Superiority; p = 0.76, Regression, Cox; Hazard Ratio (HR) = 0.97, 99.1% CI 2-sided [0.73 to 1.28]
Statistical Analysis 2: Comparison: Absence of Adjuvant Temozolomide (TMZ) vs Presence of Adjuvant Temozolomide (TMZ); Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.52 to 0.79]

2. Secondary Outcome: Progression-free Survival
Description: Disease progression is defined as radiological or neurological/clinical progression (whichever occurs first); progression free survival (PFS) is the time interval between the date of randomization and the date of disease progression or death whichever occurs first. If neither event has been observed, the patient is censored at the date of the last follow up examination. Radiological progression was defined as increase of contrast enhancing area on MRI or CT scans of more than 25% as measured by two perpendicular diameters compared to the smallest measurements ever recorded for the same lesion by the same technique. The appearance of new lesions with or without contrast enhancement Neurological/clinical progression was defined as:decrease in WHO performance status,deterioration of neurological functions,appearance of signs/symptoms of increased intracranial pressure,and/or start of corticosteroid or increase of corticosteroid dosage by 50% for control of neurological symptoms.
Time Frame: from randomization till the date of disease progression or death (time till death is up to 10.9 years after patient enrollment in the study)
Population: This trial studied separately two questions 1) effect of concomitant TMZ 2) effect of adjuvant TMZ. The 4 randomized arms were combined before analysis. Absence of concomitant TMZ including Arm RT alone & Arm RT followed by adjuvant TMZ. Presence of concomitant TMZ including Arm TMZ/RT & Arm TMZ/RT followed by adjuvant TMZ. Absence of adjuvant TMZ including Arm RT alone & Arm TMZ/RT. Presence of adjuvant TMZ including Arm RT followed by adjuvant TMZ & Arm TMZ/RT followed by adjuvant TMZ
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Absence of Concomitant TMZ: Including 2 randomized arms: Arm RT alone and Arm RT followed by adjuvant TMZ
- Presence of Concomitant TMZ: Including 2 randomized arms: Arm TMZ/RT and Arm TMZ/RT followed by adjuvant TMZ
- Absence of Adjuvant TMZ: Including two randomized arms: Arm RT alone and Arm TMZ/RT
- Presence of Adjuvant TMZ: Including to 2 randomized arms: Arm RT followed by adjuvant TMZ and Arm TMZ/RT followed by adjuvant TMZ
Arm/Group | Absence of Concomitant TMZ | Presence of Concomitant TMZ | Absence of Adjuvant TMZ | Presence of Adjuvant TMZ
Number analyzed (Participants) | 375 | 376 | 377 | 374
Months | 20.9 [17.25 to 26.64] | 33.02 [23.82 to 46.06] | 19.09 [14.59 to 23.82] | 42.81 [27.83 to 56.44]
Statistical Analysis 1: Comparison: Absence of Concomitant TMZ vs Presence of Concomitant TMZ; Test type: Superiority; p = 0.11, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.72 to 1.03]
Statistical Analysis 2: Comparison: Absence of Adjuvant TMZ vs Presence of Adjuvant TMZ; Test type: Superiority; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.49 to 0.70]

3. Secondary Outcome: Quality of Life of the Patient
Description: Quality of life was assessed by the EORTC Quality of Life Questionnaire (QLQ-C30) version 3 and the Brain Cancer Module-20
Time Frame: from 14 days prior to randomization till five years or death (time till death is up to 10.9 years after patient enrollment in the study)
Reporting Status: Not Posted, anticipated posting 2025-04

4. Secondary Outcome: Neurological Deterioration Free Survival
Description: Neurological deterioration is defined as a decrease in WHO performance status as follows:
  decrease in WHO performance status
  * for patients with baseline WHO performance status 0: deterioration to WHO performance status 2 or worse for which no other explanation is present, and which is maintained for at least three months
  * for patients with baseline WHO performance status 1 or 2: deterioration to WHO performance status 3 or worse for which no other explanation is present and which is maintained for at least three months
  The date of neurological deterioration will be the first date the persistent decrease in performance status was diagnosed. Neurological deterioration free progression is the time interval between the date of randomization and the date of neurological deterioration or death whichever occurs first. If neither event has been observed, the patient is censored at the date of the last follow up examination
Time Frame: within 2 weeks of randomization; during radiotherapy at week 4 and 6; 4 weeks after the end of radiotherapy; Six monthly after the end of radiotherapy; Prior to each cycle of adjuvant therapy; Every six months after the documentation of first progression.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of radiotherapy up to 14.5 months after patient enrolment in the study. All-Cause Mortality was assessed through study completion, up to 10.9 years after patient enrolment in the study.
Description: Both serious and non-serious AEs were collected. We reported SAEs and all AEs. Non serious AEs are accounted for in the all AEs report. All AEs report is included in the Other (Not Including Serious) section. All-cause mortality was assessed in the intent to treat population defined as all randomized patients. SAEs and all AEs were assessed in the randomized patients who have started their allocated treatments
Arm/Group | RT Alone | RT & Concurrent CT | RT + Adjuvant CT | RT & Concurrent CT + Adjuvant CT
All-Cause Mortality (participants affected / at risk) | 107/189 | 97/188 | 78/186 | 74/188
Serious Adverse Events (participants affected / at risk) | 13/186 | 27/185 | 32/183 | 32/185
Other Adverse Events (participants affected / at risk) | 182/186 | 183/185 | 182/183 | 185/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RT Alone (N=186) | RT & Concurrent CT (N=185) | RT + Adjuvant CT (N=183) | RT & Concurrent CT + Adjuvant CT (N=185)
VASCULAR (Vascular disorders) | 0 | 1 | 1 | 0
ALLERGY/IMMUNOLOGY (Immune system disorders) | 0 | 0 | 2 | 2
CONSTITUTIONAL SYMPTOMS (General disorders) | 0 | 7 | 2 | 2
PAIN (General disorders) | 2 | 2 | 4 | 3
CARDIAC(GENERAL) (Cardiac disorders) | 1 | 0 | 0 | 1
BLOOD (Blood and lymphatic system disorders) | 2 | 2 | 2 | 5
LYMPHATICS (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
PULMONARY/UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
NEUROLOGY (Nervous system disorders) | 9 | 15 | 12 | 10
OCULAR/VISUAL (Eye disorders) | 0 | 2 | 0 | 1
GASTROINTESTINAL (Gastrointestinal disorders) | 1 | 2 | 4 | 5
RENAL/GENITOURINARY (Renal and urinary disorders) | 0 | 0 | 1 | 1
DERMATOLOGY/SKIN (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 2
MUSCULOSKELETAL/SOFT TISSUE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
METABOLIC/LABORATORY (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
INFECTION (Infections and infestations) | 6 | 4 | 8 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RT Alone (N=186) | RT & Concurrent CT (N=185) | RT + Adjuvant CT (N=183) | RT & Concurrent CT + Adjuvant CT (N=185)
VASCULAR (Vascular disorders) | 2 | 7 | 5 | 7
SURGERY/INTRA-OPERATIVE INJURY (Surgical and medical procedures) | 0 | 0 | 0 | 0
ALLERGY/IMMUNOLOGY (Immune system disorders) | 7 | 9 | 11 | 9
CONSTITUTIONAL SYMPTOMS (General disorders) | 151 | 160 | 170 | 160
PAIN (General disorders) | 129 | 131 | 138 | 131
SEXUAL/REPRODUCTIVE FUNCTION (Reproductive system and breast disorders) | 2 | 4 | 7 | 4
CARDIAC(GENERAL) (Cardiac disorders) | 9 | 15 | 17 | 15
PULMONARY/UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 17 | 9
BLOOD (Blood and lymphatic system disorders) | 5 | 12 | 10 | 12
LYMPHATICS (Blood and lymphatic system disorders) | 12 | 10 | 14 | 10
NEUROLOGY (Nervous system disorders) | 147 | 153 | 148 | 153
OCULAR/VISUAL (Eye disorders) | 51 | 62 | 48 | 62
AUDITORY/EAR (Ear and labyrinth disorders) | 30 | 23 | 33 | 23
GASTROINTESTINAL (Gastrointestinal disorders) | 107 | 136 | 158 | 136
RENAL/GENITOURINARY (Renal and urinary disorders) | 11 | 7 | 16 | 7
HEPATOBILIAR/PANCREAS (Hepatobiliary disorders) | 0 | 0 | 0 | 0
DERMATOLOGY/SKIN (Skin and subcutaneous tissue disorders) | 146 | 139 | 147 | 139
MUSCULOSKELETAL/SOFT TISSUE (Musculoskeletal and connective tissue disorders) | 16 | 17 | 23 | 17
ENDOCRINE (Endocrine disorders) | 6 | 8 | 9 | 8
METABOLIC/LABORATORY (Metabolism and nutrition disorders) | 7 | 7 | 8 | 7
INFECTION (Infections and infestations) | 37 | 35 | 72 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT00626990/Prot_SAP_000.pdf